CLINICAL TRIAL: NCT00620321
Title: An Open-Label Phase 2 Trial of LY2181308 Sodium Administered in Combination With Idarubicin and Cytarabine to Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: A Study of LY2181308 Sodium in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11631; H8Z-MC-JACU (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-02-04; First posted 2008-02-21 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2181308 sodium, idarubicin, cytarabine (Experimental)
  Interventions: Drug: LY2181308 sodium; Drug: cytarabine; Drug: idarubicin

INTERVENTIONS:
Drug: LY2181308 sodium — 750 milligrams (mg) is administered as a 3-hour intravenous infusion on Days 1, 2, 3, 8, 15, 22 of Cycle 1 (28 days) and Days 1, 8, 15, 22 of Cycle 2 (28 days) until disease progression or unacceptable toxicity develops.
Drug: cytarabine — 1.5 grams per square meter (g/m²) will be administered as a 4-hour intravenous infusion on Days 3, 4, 5 of Cycle 1 (28 days) and Days 1, 2, 3 of Cycle 2 (28 days) until disease progression or unacceptable toxicity develops.
Drug: idarubicin — 12 milligrams per square meter (mg/m²) will be administered as a 30-minute intravenous infusion on Days 3, 4, 5 of Cycle 1 (28 days) and on Days 1, 2, 3 of Cycle 2 (28 days) until disease progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to understand the safety profile of LY2181308 sodium administered in combination with idarubicin and cytarabine to patients with relapsed or refractory acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of acute myeloid leukemia that is relapsed or refractory to at least 1 prior treatment for leukemia, or patients with chronic myeloid leukemia (CML) who are in myeloid blast crisis which have failed at least 1 previous tyrosine kinase inhibitor (TK1). A baseline bone marrow assessment is required less than or equal to 96 hours prior to the first dose of study drug.
* Must have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, immunotherapy, cancer related hormone therapy, or other investigational therapy for at least 21 days for myelosuppressive agents (such as cytarabine, daunorubicin, and gemtuzumab ozogamicin) or 14 days for non-myelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy (such as neurotoxicity, diarrhea, and mucositis) except for residual myelosuppression and alopecia. Hydroxyurea is permitted to control the peripheral blast cell count, but must be stopped at least 24 hours before study drug administration.
* Must have adequate organ function.
* Females must have a negative pregnancy test. Male and female patients must agree to use a reliable method of birth control during and for 6 months following the last dose of study drug.
* Patients must be at least 18 years old.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a non-myelosuppressive or myelosuppressive agent, respectively.
* Patients with acute promyelocytic leukemia (APML).
* Major surgery within 4 weeks of study enrollment.
* Patients with serious pre-existing medical conditions (at the discretion of the investigator). Because of the known cardiac toxicity of anthracyclines, patients with pre-existing ejection fraction (EF) less than or equal to 45% should not participate in this study. No patient should exceed the maximum exposure of anthracycline doses (for example, idarubicin greater than 120 mg/m²).
* Patients with a second malignancy that could affect the interpretation of the results.
* Patients with leukemic involvement of the central nervous system (CNS) by spinal fluid cytology or imaging.
* Patients with known coagulopathy or bleeding disorder, other than leukemia related thrombocytopenia. Patients with severe of life threatening bleeding refractory to platelet transfusions are also excluded.
* Concomitant anticoagulant therapy (with the exception of heparinized saline to maintain the patency of central venous catheters).
* Women who are pregnant or breast feeding.
* Patients with a known hypersensitivity to oligonucleotides, idarubicin, and/or cytarabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Erba HP, Sayar H, Juckett M, Lahn M, Andre V, Callies S, Schmidt S, Kadam S, Brandt JT, Van Bockstaele D, Andreeff M. Safety and pharmacokinetics of the antisense oligonucleotide (ASO) LY2181308 as a single-agent or in combination with idarubicin and cytarabine in patients with refractory or relapsed acute myeloid leukemia (AML). Invest New Drugs. 2013 Aug;31(4):1023-34. doi: 10.1007/s10637-013-9935-x. Epub 2013 Feb 10. PMID 23397500
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the Participant Flow are the reasons the participant discontinued treatment. All participants who have completed at least 1 cycle of study drug were considered to have completed the study.
Groups:
- LY2181308: 750 milligrams (mg) was administered as a 3-hour intravenous infusion on Days 1, 2, 3, 8, 15, 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycle 2 and beyond. Cycle length: 28 days.
- LY2181308 + Idarubicin + Cytarabine: LY2181308: 750 mg was administered as a 3-hour intravenous infusion on Days 1, 2, 3, 8, 15, 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycle 2 and beyond.
  Idarubicin: 12 milligrams per square meter (mg/m²) was administered as a 30-minute intravenous infusion on Days 3, 4, 5 of Cycle 1 and on Days 1, 2, 3 of Cycle 2 and beyond.
  Cytarabine: 1.5 grams per square meter (g/m²) was administered as a 4-hour intravenous infusion on Days 3, 4, 5 of Cycle 1 and Days 1, 2, 3 of Cycle 2 and beyond.
  Cycle length: 28 days.
Period: Overall Study
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Started | 8 | 16
Received at Least 1 Dose of Study Drug | 8 | 16
Completed | 0 | 0
Not Completed | 8 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 1
Not completed — Physician Decision | 0 | 7
Not completed — Progressive Disease | 5 | 5
Not completed — Sponsor Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine | Total
Number analyzed (Participants) | 8 | 16 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.26 (15.93) | 48.22 (14.72) | 52.23 (15.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 3 | 10 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 0 | 2 | 2
  Caucasian | 7 | 11 | 18
  East Asian | 1 | 0 | 1
  Hispanic | 0 | 1 | 1
  West Asian | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (Safety Profile)
Description: Data are presented as number of participants who experienced serious adverse events (SAE) and possibly drug-related treatment-emergent adverse events (TEAE) during the study including the 21-day follow-up period. A summary of serious adverse events and other nonserious adverse events regardless of causality is located in the Reported Adverse Events section.
Time Frame: Start of treatment to study completion up to 6.7 months
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Number analyzed (Participants) | 8 | 16
Participants
  SAE | 6 | 13
  Drug-related TEAE | 2 | 11

2. Secondary Outcome: Percentage of Participants With Response to LY2181308 Sodium in Combination With Idarubicin and Cytarabine (Remission Rates)
Description: Response is complete remission (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) + cytoreduction. CR: fewer than 5% blasts based on a cell count of at least 200 cells from a bone marrow aspirate containing bone marrow spicules, in the setting of peripheral blood recovery to: platelets ≥100x10⁹/liter (L), neutrophils ≥10⁹/L. PR: defined as a decrease of at least 50% in blast count on the bone marrow aspirate; or cytoreduction (defined as a decrease in blast count not meeting the criteria for a PR or CR). Response rate is calculated as a total number of participants with CR or CRi or PR or cytoreduction divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline to progression of disease or death up to 6 months
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Number analyzed (Participants) | 8 | 16
percentage of participants | 0 | 56.3

3. Secondary Outcome: Relapse-Free Survival
Description: Relapse-Free Survival was defined as the time from first objective status assessment of complete remission (CR) or CR with incomplete blood count recovery (CRi) or partial remission (PR) or cytoreduction to the first time of disease progression or death as a result of any cause. CR: fewer than 5% blasts based on a cell count of at least 200 cells from a bone marrow aspirate containing bone marrow spicules, in the setting of peripheral blood recovery to: platelets ≥100x10⁹/liter (L), neutrophils ≥10⁹/L. PR: defined as a decrease of at least 50% in blast count on the bone marrow aspirate; or cytoreduction (defined as a decrease in blast count not meeting the criteria for a PR or CR). There were too few participants who had a documented progression of disease or death event amongst the participants with a response of CR, CRi, PR or cytoreduction to conduct the time-to-event analysis, thus the relapse-free survival was not analyzed.
Time Frame: Baseline to progression of disease or death up to 6 months
Population: Zero participants analyzed as no data collected on participants for relapse free survival due to no sufficient follow up on participants with response for time to event.
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Area Under the Curve of LY2181308 Over the Dosing Interval
Description: Area under the curve of LY2181308 over the dosing interval
Time Frame: Day 3: 0,12,24,36,48,60,72,84,96,108,120,132 hours
Population: All participants who received study drug and had pharmacokinetic (PK) data to calculate AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Number analyzed (Participants) | 8 | 16
nanograms*hour/milliliter (ng*h/mL) | 216947 (60.0) | 185734 (45.7)

5. Secondary Outcome: Pharmacodynamics: Number of Participants With Survivin Protein Expression
Description: Pharmacodynamics: Number of participants with Survivin Protein Expression.
Time Frame: 6 Months
Population: All participants who received at least one dose of study drug. Per protocol amendment, Survivin Protein Expression change was assessed for LY2181308 arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2181308
Number analyzed (Participants) | 8
Participants | 2

6. Secondary Outcome: Change From Baseline in Survivin Index at Day 2
Description: Data presented are the ratio of Day 2 survivin index to the baseline survivin index. Survivin is a protein expressed in tumor cells, including acute myeloid leukemia (AML), which regulates mitosis and prevents tumor cell death. Survivin index was calculated as ([blast survivin mean equivalent fluorochrome (MEFL) - blast isotypic control MEFL]/blast isotypic control MEFL).
Time Frame: Baseline, Day 2
Population: All participants who received at least one dose of study drug and had both baseline and Day 2 survivin index measurements. Per protocol amendment, only participants in LY2181308 arm were analyzed for Survivin Index.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | LY2181308
Number analyzed (Participants) | 8
ratio | 0.43 [0.28 to 0.67]

7. Other Pre Specified Outcome: Number of Participants Who Died Due to Progressive Disease or Unknown Cause During the 21 Days Post Study Treatment Follow-Up
Description: Deaths due to progressive disease (PD) and unknown cause are not considered adverse events. Deaths due to PD and unknown cause occurring during the 21-day follow-up period after treatment discontinuation are reported here and for those occurring while participants were on treatment are reported in the Participant Flow. Deaths due to serious adverse events occurred during the study including the 21-day follow-up period are reported in the Reported Adverse Events section.
Time Frame: Study treatment discontinuation up to 21 days post study treatment discontinuation
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Number analyzed (Participants) | 8 | 16
Participants
  Death due to progressive disease | 1 | 0
  Death due to unknown cause | 1 | 0

ADVERSE EVENTS:
Description: Deaths due to progressive disease and unknown cause are not considered adverse events and are reported in the Participant Flow for those participants who died while taking study drug. Deaths due to progressive disease or unknown cause during the 21-day post-study treatment follow-up period are reported in the Other Pre-Specified Outcome Measure.
Arm/Group | LY2181308 | LY2181308 + Idarubicin + Cytarabine
Serious Adverse Events (participants affected / at risk) | 6/8 | 13/16
Other Adverse Events (participants affected / at risk) | 8/8 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2181308 (N=8) | LY2181308 + Idarubicin + Cytarabine (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 0 (0) | 1 (1) — Event resulted in 1 death in the LY2181308+Cytarabine+Idarubicin arm during the post-therapy follow-up period.
Clostridial infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) — Event resulted in 1 death in the LY2181308 arm during the treatment period.
Sepsis (Infections and infestations) | 4 (4) | 1 (1) — Event resulted in 3 deaths in the LY2181308 arm during the post-therapy follow-up period.
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Event resulted in 2 deaths in the LY2181308+Cytarabine+Idarubicin arm; 1 death during the treatment period and 1 death during the post-therapy follow-up period.
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2181308 (N=8) | LY2181308 + Idarubicin + Cytarabine (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (5)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (7)
Abdominal rebound tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (8)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Asthenia (General disorders) | 3 (3) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 6 (6)
Crepitations (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 4 (5)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 3 (6)
Pain (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Glomerular filtration rate (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (3)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (4)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 5 (5)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/5 (0) | 1/6 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (8)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 5 (6)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days